CLINICAL TRIAL: NCT05278871
Title: A Pilot Study of Noninvasive Assessment of Lymphedema Among Breast Cancer Survivors
Brief Title: Noninvasive Assessment of Lymphedema Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microelastic Ultrasound Systems Inc (Industry)
Collaborators: Duke Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00109917
Record Dates: First submitted 2022-02-28; First posted 2022-03-14 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Lymphedema of Upper Arm; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CSI ultrasound measurement (Experimental): Participants will have standard volumetric tape measurement across multiple arm locations for lymphedema followed by CSI ultrasound measurements of the same anatomic sites.
  Interventions: Device: Constructive Shearwave Interference (CSI)

INTERVENTIONS:
Device: Constructive Shearwave Interference (CSI) — handheld ultrasound
  Other Names: Bullseye Elasticity Quantification

SUMMARY:
This proof of concept study will evaluate the ability of a new, ultrasound based technology called Bullseye Constructive Shearwave Interference (CSI) (trade name, Bullseye Elasticity Quantification) to measure lymphedema of the upper arm among breast cancer survivors.

The study's hypothesis is that the CSI device can detect the presence of clinically significant lymphedema when compared with the standard arm tape measurement.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with a history of unilateral breast cancer who has completed definitive treatment for breast cancer (i.e. previously undergone surgical resection, with or without adjuvant radiotherapy and/or chemotherapy). Subjects must have completed all recommended adjuvant radiotherapy. Subjects who continue on systemic therapy may be included at the discretion of the treating physician.
* Subjects with a history of unilateral axillary sentinel biopsy, lymphadenectomy or dissection are eligible for inclusion.
* Subjects taking hormonal therapy are eligible for inclusion
* Subject has any stage lymphedema

Exclusion Criteria:

* Active rash or skin tears/injury in bilateral upper extremities
* Subjects with history of contralateral breast cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Difference in mean shear wave speed across sites measured between lymphedema and non-lymphedema limbs | baseline
  differences in shear wave speed (Bullseye) device measurements between lymphedema affected and non-affected contralateral limb

CONTACTS AND LOCATIONS:
Overall Officials: Susan McDuff, MD PhD, Principal Investigator — Duke Health
Locations (2):
- United States (2):
  - Durham Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SY, Cardones AR, Doherty J, Nightingale K, Palmeri M. Preliminary Results on the Feasibility of Using ARFI/SWEI to Assess Cutaneous Sclerotic Diseases. Ultrasound Med Biol. 2015 Nov;41(11):2806-19. doi: 10.1016/j.ultrasmedbio.2015.06.007. Epub 2015 Aug 8. PMID 26259888